CLINICAL TRIAL: NCT01271452
Title: Safety and Efficacy of Two Types of Botulinum Toxin Type A For the Treatment of Glabellar Lines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAF/AGN/Facial/011; 2010-021401-20 (EudraCT Number)
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Results first posted 2012-01-16 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Glabellar Lines
MeSH Terms: interventions — Botulinum Toxins, Type A; incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vistabel® (Active Comparator): botulinum toxin type A (Vistabel®)
  Interventions: Biological: botulinum toxin type A
- Bocouture® (Active Comparator): botulinum toxin type A (Bocouture®)
  Interventions: Biological: botulinum toxin type A

INTERVENTIONS:
Biological: botulinum toxin type A — 20 units (total dose) botulinum toxin type A injected into glabellar region on Day 0
  Other Names: Vistabel®; BOTOX® Cosmetic
  Arms: Vistabel®
Biological: botulinum toxin type A — 30 units (total dose) botulinum toxin type A injected into glabellar region on Day 0
  Other Names: Bocouture®
  Arms: Bocouture®

SUMMARY:
This study will evaluate the safety and efficacy of two different types of botulinum toxin type A for the treatment of glabellar frown lines.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe glabellar frown lines

Exclusion Criteria:

* Diagnosis of myasthenia gravis or Eaton Lambert syndrome
* Aesthetic treatment with botulinum toxin within 6 months or planned treatment with botulinum toxin for any reason during the study
* Prior filler treatments, surgeries, insertion procedures in/to the glabellar region
* Facial cosmetic procedures in the glabellar area within 6 months
* Bleeding disorders or use of anticoagulants within 10 days
* History of facial nerve palsy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2010-09; Primary Completion 2011-01 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Munich, Bavaria, Germany

REFERENCES:
- [Background] Moers-Carpi M, Dirschka T, Feller-Heppt G, Hilton S, Hoffmann K, Philipp-Dormston WG, Rutter A, Tan K, Chapman MA, Fulford-Smith A. A randomised, double-blind comparison of 20 units of onabotulinumtoxinA with 30 units of incobotulinumtoxinA for glabellar lines. J Cosmet Laser Ther. 2012 Dec;14(6):296-303. doi: 10.3109/14764172.2012.738913. Epub 2012 Nov 15. PMID 23057624

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vistabel® | Bocouture®
Started | 112 | 112
Completed | 105 | 104
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vistabel® | Bocouture® | Total
Number analyzed (Participants) | 112 | 112 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (10.80) | 45.4 (9.82) | 45.2 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 102 | 200
  Male | 14 | 10 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With a Treatment Response at Day 28 Based on the Injector's Assessment of the Severity of Glabellar Lines at Maximum Contraction Using the Facial Wrinkle Scale (FWS)
Description: Number of subjects with a treatment response at Day 28 based on the injector's assessment of the severity of glabellar lines at maximum contraction using the FWS. The FWS measures wrinkles on a scale from 0=none (best) to 3=severe (worst). Treatment response was defined as a 1 point or greater reduction from Day 0 in the FWS score at maximum contraction.
Time Frame: Day 28
Population: Intent-to-treat (ITT): all randomized subjects.
Measure: Number; unit: Number of Subjects
Arm/Group | Vistabel® | Bocouture®
Number analyzed (Participants) | 112 | 112
Number of Subjects | 108 | 106

2. Secondary Outcome: Number of Subjects With a Treatment Response at Day 84 Based on the Injector's Assessment of the Severity of Glabellar Lines at Maximum Contraction Using the FWS
Description: Number of subjects with a treatment response at Day 84 based on the injector's assessment of the severity of glabellar lines at maximum contraction using the FWS. The FWS measures wrinkles on a scale from 0=none (best) to 3=severe (worst). Treatment response was defined as a 1 point or greater reduction from Day 0 in the FWS score at maximum contraction.
Time Frame: Day 84
Population: ITT: all randomized subjects.
Measure: Number; unit: Number of Subjects
Arm/Group | Vistabel® | Bocouture®
Number analyzed (Participants) | 112 | 112
Number of Subjects | 90 | 80

3. Secondary Outcome: Number of Subjects With a Treatment Response at Day 98 Based on the Injector's Assessment of the Severity of Glabellar Lines at Maximum Contraction Using the FWS
Description: Number of subjects with a treatment response at Day 98 based on the injector's assessment of the severity of glabellar lines at maximum contraction using the FWS. The FWS measures wrinkles on a scale from 0=none (best) to 3=severe (worst). Treatment response was defined as a 1 point or greater reduction from Day 0 in the FWS score at maximum contraction.
Time Frame: Day 98
Population: ITT: all randomized subjects.
Measure: Number; unit: Number of Subjects
Arm/Group | Vistabel® | Bocouture®
Number analyzed (Participants) | 112 | 112
Number of Subjects | 76 | 70

4. Secondary Outcome: Number of Subjects With a Treatment Response at Day 112 Based on the Injector's Assessment of the Severity of Glabellar Lines at Maximum Contraction Using the FWS
Description: Number of subjects with a treatment response at Day 112 based on the injector's assessment of the severity of glabellar lines at maximum contraction using the FWS. The FWS measures wrinkles on a scale from 0=none (best) to 3=severe (worst). Treatment response was defined as a 1 point or greater reduction from Day 0 in the FWS score at maximum contraction.
Time Frame: Day 112
Population: ITT: all randomized subjects.
Measure: Number; unit: Number of Subjects
Arm/Group | Vistabel® | Bocouture®
Number analyzed (Participants) | 112 | 112
Number of Subjects | 61 | 56

5. Secondary Outcome: Number of Subjects With a Treatment Response at Day 28 Based on the Subject's Assessment of the Severity of Glabellar Lines at Maximum Contraction Using the FWS
Description: Number of subjects with a treatment response at Day 28 based on the subject's assessment of the severity of glabellar lines at maximum contraction using the FWS. The FWS measures wrinkles on a scale from 0=none (best) to 3=severe (worst). Treatment response was defined as a 1 point or greater reduction from Day 0 in the FWS score at maximum contraction.
Time Frame: Day 28
Population: ITT: all randomized subjects.
Measure: Number; unit: Number of Subjects
Arm/Group | Vistabel® | Bocouture®
Number analyzed (Participants) | 112 | 112
Number of Subjects | 108 | 102

6. Secondary Outcome: Number of Subjects With a Treatment Response at Day 84 Based on the Subject's Assessment of the Severity of Glabellar Lines at Maximum Contraction Using the FWS
Description: Number of subjects with a treatment response at Day 84 based on the subject's assessment of the severity of glabellar lines at maximum contraction using the FWS. The FWS measures wrinkles on a scale from 0=none (best) to 3=severe (worst). Treatment response was defined as a 1 point or greater reduction from Day 0 in the FWS score at maximum contraction.
Time Frame: Day 84
Population: ITT: all randomized subjects.
Measure: Number; unit: Number of Subjects
Arm/Group | Vistabel® | Bocouture®
Number analyzed (Participants) | 112 | 112
Number of Subjects | 84 | 78

7. Secondary Outcome: Number of Subjects With a Treatment Response at Day 98 Based on the Subject's Assessment of the Severity of Glabellar Lines at Maximum Contraction Using the FWS
Description: Number of subjects with a treatment response at Day 98 based on the subject's assessment of the severity of glabellar lines at maximum contraction using the FWS. The FWS measures wrinkles on a scale from 0=none (best) to 3=severe (worst). Treatment response was defined as a 1 point or greater reduction from Day 0 in the FWS score at maximum contraction.
Time Frame: Day 98
Population: ITT: all randomized subjects.
Measure: Number; unit: Number of Subjects
Arm/Group | Vistabel® | Bocouture®
Number analyzed (Participants) | 112 | 112
Number of Subjects | 73 | 68

8. Secondary Outcome: Number of Subjects With a Treatment Response at Day 112 Based on the Subject's Assessment of the Severity of Glabellar Lines at Maximum Contraction Using the FWS
Description: Number of subjects with a treatment response at Day 112 based on the subject's assessment of the severity of glabellar lines at maximum contraction using the FWS. The FWS measures wrinkles on a scale from 0=none (best) to 3=severe (worst). Treatment response was defined as a 1 point or greater reduction from Day 0 in the FWS score at maximum contraction.
Time Frame: Day 112
Population: ITT: all randomized subjects.
Measure: Number; unit: Number of Subjects
Arm/Group | Vistabel® | Bocouture®
Number analyzed (Participants) | 112 | 112
Number of Subjects | 61 | 54

ADVERSE EVENTS:
Description: The Safety Population was used to analyze serious adverse events and adverse events and consisted of all randomised subjects who received at least one administration of study treatment (to at least one injection site). One subject in the Bocouture® treatment group was not included in the Safety Population.
Arm/Group | Vistabel® | Bocouture®
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/111
Other Adverse Events (participants affected / at risk) | 6/112 | 2/111
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vistabel® (N=112) | Bocouture® (N=111)
Nasopharyngitis (Infections and infestations) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is at least 30 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication and can extend the embargo